CLINICAL TRIAL: NCT00553293
Title: Recombinant LH Supplementation to Recombinant FSH During the Final Days of Controlled Ovarian Stimulation for IVF: a Multicentre, Prospective, Randomized, Controlled Trial
Brief Title: Nordic Luveris Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Regionshospitalet Viborg, Skive (Other); Karolinska University Hospital (Other); Helse Fonna (Other); Turku Hospital (Unknown); Odense University Hospital (Other); Herlev Hospital (Other); Holbaek Sygehus (Other); Hvidovre University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KF02-035/03
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Infertility; In Vitro Fertilization
Keywords: infertility; in vitro fertilization; LH supplementation; Benefits
MeSH Terms: conditions — Infertility | interventions — Luteinizing Hormone; Luteinizing Hormone, beta Subunit; Glycoprotein Hormones, alpha Subunit; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A,1 (Active Comparator): rFSH + rLH arm
  Interventions: Drug: recombinant luteinizing hormone (Luveris)
- A,2 (Placebo Comparator): rFSH alone
  Interventions: Drug: recombinant follicle stimulating hormone (Gonal-f)

INTERVENTIONS:
Drug: recombinant luteinizing hormone (Luveris) — 75 iu/day form cycle day 6
  Other Names: Luveris
  Arms: A,1
Drug: recombinant follicle stimulating hormone (Gonal-f) — rFSH 150 iu/day
  Other Names: Gonal-f
  Arms: A,2

SUMMARY:
To study whether addition of human LH hormone (Luveris) during the final days of stimulation with recombinant FSH (Gonal-f) for controlled ovarian stimulation will be of benefit for patients undergoing in vitro fertilisation.

ELIGIBILITY:
Inclusion Criteria:

* Age below 40
* Infertility treatable by IVF or ICSI
* Regular cycles

Exclusion Criteria:

* NA

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 526 (Actual)
Dates: Start 2003-08; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate per started stimulation cycle | ultrasound showing ongoing pregnancy

SECONDARY OUTCOMES:
Ongoing pregnancy in subgroups of patients with lo0w serum LH levels | ultrasound for ongoing pregnancy in subgroups

CONTACTS AND LOCATIONS:
Overall Officials: Anders N Andersen, professor, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Anders Nyboe Andersen, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] NyboeAndersen A, Humaidan P, Fried G, Hausken J, Antila L, Bangsboll S, Rasmussen PE, Lindenberg S, Bredkjaer HE, Meinertz H; Nordic LH study group. Recombinant LH supplementation to recombinant FSH during the final days of controlled ovarian stimulation for in vitro fertilization. A multicentre, prospective, randomized, controlled trial. Hum Reprod. 2008 Feb;23(2):427-34. doi: 10.1093/humrep/dem317. Epub 2007 Nov 16. PMID 18024487